CLINICAL TRIAL: NCT05972668
Title: Smartphone App for Asthma Self-care: Assessment of Outcomes (Asthma Progession and Costs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Collaborators: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, I-Jen, Wang, Clinical Professor, Taipei Hospital, Ministry of Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TH-IRB-0016-0038
Record Dates: First submitted 2023-07-07; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: Smartphone selft-care system; asthma control; medical cost; emergency room visit; hospital admission
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group needs to download the smartphone apps and follow research protocol
  Interventions: Device: Smartphone Apps
- Control group (No Intervention)

INTERVENTIONS:
Device: Smartphone Apps — The intervention group downloaded the asthma smartphone app, and followed up monthly via phone calls and clinic visits
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to investigate whether a smartphone app based on the Global Initiative for Asthma (GINA) guidelines can improve asthma control and quality of life, and decrease asthma-related costs in children. The main question it to answer whether this app can improve asthma control, increase the quality of life, and decrease asthma-related costs.

Participants in the intervention group downloaded the asthma smartphone app, and followed up monthly via phone calls and clinic visits, while the control group received reminder calls. Researchers will compare with the control group to see if the intervention receives more asthma control improvement.

ELIGIBILITY:
Inclusion Criteria:

* aged between 3 and 18 years;
* who had access to the smartphone app;
* with asthma treatment steps 2-4, requiring regular treatment with controller medication (for at least 6 months over the past year) according to the GINA guidelines;
* who had at least two clinic or emergency department visits related to asthma in the previous year.

Exclusion Criteria:

* Children who had comorbidities, or other major medical problems, and who did not have a smartphone or whose caregivers did not have a smartphone were excluded from the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants both in intervention and control were assessed for the asthma severity change using Global Strategy for Asthma Management and Prevention (GINA) Guideline | 3 and 6 months evaluation
  The physician diagnoses asthma change at Taipei Hospital
All participants were assessed for the Asthma Control Test (ACT) change using ACT questionnaire from quality metric incorporated | 3 and 6 months evaluation
  The physician evaluate ACT change at Taipei Hospital for both group
All participants were assessed for the change of Quality of life using MiniPAQLQ | 3 and 6 months evaluation
  Physician and researchers evaluate the quality of life using MiniPAQLQ questionnaire
All participants were assessed for the Asthma Control Test change using Paediatric Asthma Quality of Life Questionnaire (PAQLQ) questionnaire | 3 and 6 months evaluation
  The physician evaluate PASS score change at Taipei Hospital for both group
All participants were assessed for the Peak Expiratory Flow (PEF) change using spirometry | 3 and 6 months
  The physician evaluate PEF change at Taipei Hospital for both group
All participants were assessed for the change of asthma cost using direct and indirect costs from national website | 3 and 6 months
  Researchers access the data from National Health Insurance database

SECONDARY OUTCOMES:
All participants were assessed for their age in the baseline using data of birthday information | Baseline
  Nurses and or researchers is responsible in filling the data from the patient admission in the Hospital
All participants were assessed for the total serum IgE (kU/I) change from blood assessment | 3 and 6 months evaluation
  The researcher and physician record and evaluate the data
All participants were assessed for the comorbidities with atopic dermatitis using the health data record from Hospital and National Health Insurance | Baseline
  The researcher and physician record and evaluate the data
All participants were assessed for the comorbidities with allergic rhinitis using the health data record from Hospital and National Health Insurance | Baseline
  The researcher and physician record and evaluate the data
All participants were assessed for the family history of atopic disease using the health data record from Hospital and National Health Insurance | Baseline
  The researcher and physician record and evaluate the data
All participants were assessed for the systemic steroid dosage (prednisolone, mg), using the health data record from Hospital and National Health Insurance | Baseline
  The researcher and physician record and evaluate the data
All participants were assessed for the ICS Dosage (Seretide,mcg), using the health data record from Hospital and National Health Insurance | Baseline
  The researcher and physician record and evaluate the data
All participants were assessed for the Anti-leukotriene (montelukast, tab), using the health data record from Hospital and National Health Insurance | Baseline
  The researcher and physician record and evaluate the data

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
We don not plan to share individual participant data (IPD)

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT05972668/SAP_000.pdf